CLINICAL TRIAL: NCT04273672
Title: Speech, Linguistic and Acoustic Markers in Parkinson's Disease
Acronym: SLAM-PD
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Boston University (Other); VA Puget Sound Health Care System (U.S. Federal Agency); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Massachusetts Institute of Technology/Lincoln Labs (Unknown)
Responsible Party: Principal Investigator, Kara Smith, Assistant Professor of Neurology, University of Massachusetts, Worcester
Other Study IDs: H00011523; 5K23DC016656 (NIH)
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Cognitive Impairment, Mild; Speech
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Speech | interventions — Voice; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease: Subjects with Parkinson's Disease
  Interventions: Diagnostic Test: Cognitive Battery; Behavioral: Voice, Speech and Language Analysis; Behavioral: Questionnaires and Clinical Assessments; Genetic: DNA Analysis
- Control: Subjects without Parkinson's Disease
  Interventions: Diagnostic Test: Cognitive Battery; Behavioral: Voice, Speech and Language Analysis; Behavioral: Questionnaires and Clinical Assessments

INTERVENTIONS:
Diagnostic Test: Cognitive Battery — Participants will be asked to complete a series of cognitive testing (testing of concentration, memory, and other thinking abilities).
Behavioral: Voice, Speech and Language Analysis — Participants will be asked to perform speaking and reading tasks, which will be recorded. Participants will be asked to complete a laptop-based test of language comprehension.
Behavioral: Questionnaires and Clinical Assessments — Participants with Parkinson's disease will complete an examination of their symptoms and questionnaires assessing disease symptoms, mood and activities of daily living. Healthy controls participants will be asked to complete questionnaires on mood.
Genetic: DNA Analysis — Participants will have their blood drawn for DNA analysis.
  Groups: Parkinson's Disease

SUMMARY:
The Investigators aim to identify speech and language markers that provide information on cognitive function and predict cognitive decline in Parkinson's disease. The Investigators will administer speech tasks and cognitive assessments to participants with Parkinson's disease and healthy controls. The Investigators will also explore the associations between genetic factors and speech and cognitive status in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease (or healthy control)
* Disease duration ≥ 2 years
* Mild cognitive impairment or normal cognition

Exclusion Criteria:

* Diagnosis of dementia (MoCA <21)
* Adults unable to consent
* Age < 18
* Pregnant women
* Prisoners
* Non-English speakers
* Any neurological disorder other than PD
* Deep brain stimulator placement
* Severe, unstable psychiatric disorder
* Unintelligible speech due to effects of PD
* Visual acuity or color vision impairment that would interfere with cognitive testing
* Other voice, speech or swallowing disorders or history of surgery involving palate/nasopharynx/larynx/vocal cords

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with Parkinson's Disease and mild cognitive impairment or normal cognition as well as controls
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Smith, MD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School/UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Parkinson's Disease: Participants with Parkinson's Disease with Mild Cognitive Impairment or normal cognitive function
- Control: Neurotypical controls
Period: Overall Study
Arm/Group | Parkinson's Disease | Control
Started | 49 | 9
Completed | 49 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population is the same as the assignment information, all enrolled participants were analyzed. One participant could not be appropriately categorized into the cognitive subgroups, thus the number of participants with cognitive categorization was 48.
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease | Control | Total
Number analyzed (Participants) | 49 | 9 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (7.5) | 67.0 (11.8) | 67.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 33 | 2 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 9 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 47 | 9 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mild cognitive impairment [Count of Participants; unit: Participants] — MCI in Parkinson's disease participants according to MDS Task Force Level II Criteria
  Participants | 25 | 0 | 25
Mean fundamental frequency [Mean (Standard Deviation); unit: hz] — This acoustic measure is related to average pitch of voice. It was measured using Praat software during picture description task, in all participants.
  hz | 137.9 (37.7) | 166.4 (29.7) | 142.3 (36.5)

OUTCOME MEASURES:

1. Primary Outcome: Mild Cognitive Impairment
Description: Mild cognitive impairment classified by Movement Disorders Society Task Force Level II Critieria
Time Frame: baseline
Population: The entire baseline cohort was analyzed (n=49). Per pre-specified exclusion criteria, one participant determined to have dementia (n=1) was excluded from outcome measure analysis reporting, thus the outcome measure data represents n=48 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Parkinson's Disease | Control
Number analyzed (Participants) | 49 | 9
Participants
  Parkinson's disease with mild Cognitive Impairment | 25 | 0
  Parkinson's disease with normal cognition | 23 | 9

2. Primary Outcome: Mean Fundamental Frequency
Description: These acoustic measures during spontaneous speech (picture description) were calculated using Praat
Time Frame: baseline
Population: same as enrolled
Measure: Mean (Standard Deviation); unit: Hz
Groups:
- Parkinson's Disease: Participants with Parkinson's Disease and normal cognitive status
- Parkinson's Disease With Mild Cognitive Impairment: Parkinson's disease with Mild cognitive impairment as defined by Movement disorders Society Task Force Level II critieria
- Controls: Neurotypical controls without neurological disorder
Arm/Group | Parkinson's Disease | Parkinson's Disease With Mild Cognitive Impairment | Controls
Number analyzed (Participants) | 25 | 23 | 9
Hz | 137.7 (39.6) | 142.4 (39.6) | 166.4 (29.7)

ADVERSE EVENTS:
Time Frame: This was a single visit, cross-sectional study. Adverse event data was collected during the single half-day study visit only.
Arm/Group | Parkinson's Disease | Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/9
Other Adverse Events (participants affected / at risk) | 0/49 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT04273672/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT04273672/ICF_001.pdf